CLINICAL TRIAL: NCT00200434
Title: A Double-Blind, Multi-Center, Randomized, Placebo-Controlled, Parallel Group Study of the Efficacy and Safety of Nebivolol Added to Existing Antihypertensive Treatment in Patients With Mild to Moderate Hypertension
Brief Title: A Study of the Efficacy and Safety of Nebivolol Added to Existing Antihypertensive Treatment in Patients With Hypertension
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Mylan Bertek Pharmaceuticals (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NEB321
Record Dates: First submitted 2005-09-12; First posted 2005-09-20 (Estimated); Last update posted 2005-09-20 (Estimated); Status verified 2005-09

CONDITIONS: Hypertension
Keywords: Nebivolol; Beta-Blocker; Hypertension
MeSH Terms: conditions — Hypertension | interventions — Nebivolol

INTERVENTIONS:
Drug: Nebivolol

SUMMARY:
The purpose of this study was to contrast the efficacy and safety of 3 dose levels of nebivolol vs. placebo, when added to a patient's existing antihypertensive medication(s) for 3 months, in patients with mild to moderate hypertension

DETAILED DESCRIPTION:
Following a washout of any previous beta-blocker medication, if applicable, supine, sitting, and standing cuff blood pressure and pulse rate, 24-hour ambulatory blood pressure monitoring (ABPM), ECG, laboratory assessments and genomics testing were performed before randomization. Patients were randomized to receive placebo or nebivolol once daily in the morning together with their curently prescribed antihypertensive therapy. Patients had four scheduled clinical visits during the study, following the screening visit.

ELIGIBILITY:
Inclusion Criteria:

* Average sitting diastolic blood pressure (DBP) greater then or equal to 90 mmHg and less then or equal to 109 mmHg at screening and baseline, in patients on background antihypertensive therapy taking at least one and no more than two of either ACE inhibitor, ARB, or diuretic.

Exclusion Criteria:

* Recent myocardial infarction or stroke
* Contraindications to beta-blocker therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600
Dates: Start 2002-10; Study Completion 2003-10

PRIMARY OUTCOMES:
The change from baseline to week 12 in the average sitting DBP at trough.

SECONDARY OUTCOMES:
Change from baseline to week 2, 6, and 12 in the average sitting, supine, standing systolic and diastolic blood pressure and sitting HR.

CONTACTS AND LOCATIONS:
Overall Officials: Betty S. Riggs, MD, MBA, Study Director — Mylan Pharmaceuticals Inc
Locations (1):
- Mylan Pharmaceuticals Inc., Morgantown, West Virginia, United States